CLINICAL TRIAL: NCT05580809
Title: CT Perfusion Parameters for Advanced HCC Treated by Systemic Immunotherapy : a Pilot Study
Brief Title: CT Perfusion Parameters for Advanced HCC Treated by Systemic Immunotherapy
Status: Completed | Type: Observational
Sponsor: Valérie LAURENT (Other)
Responsible Party: Sponsor-Investigator, Valérie LAURENT, MD, PhD, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2022PI117
Record Dates: First submitted 2022-10-07; First posted 2022-10-14 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Advanced HCC Treated by Systemic Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to compare CT perfusion parameters to RECIST 1.1 and mRECIST assessment for advanced HCC treated by systemic immunotherapy, and to evaluate perfusion parameters as predictive factors of response on baseline and on early follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Proved HCC
* Advanced HCC, defined as Barcelona Clinic Liver Classifications (BCLC) stage B non eligible for loco-regional therapy and stage C
* No prior systemic therapy
* Measurable disease per Response Evaluation Criteria for Solid Tumour (RECIST) v1.1
* Child-Pugh Score = A
* Eastern Cooperative Oncology Group (ECOG) Performance Status < 2

Exclusion Criteria:

* Absence of CT perfusion before treatment initiation more than a two-month delay between treatment initiation and first post-treatment CT perfusion
* Uninterpretable CT perfusion
* Definitive contraindication to CT perfusion (allergy or advanced renal disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HepatoCellular Carcinoma (HCC) treated by systemic immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Comparison of CT perfusion parameters between the responders and non-responders according to RECIST 1.1 assessment for advanced HCC treated by systemic immunotherapy | Through study completion, an average of 1 year
  Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 assessed by a senior radiologist. Comparison assessed by t test or Mann-Whitney test.
Comparison of CT perfusion parameters between the responders and non-responders according to mRECIST assessment for advanced HCC treated by systemic immunotherapy | Through study completion, an average of 1 year
  modified Response Evaluation Criteria in Solid Tumors (mRECIST) assessed by a senior radiologist. Comparison assessed by t test or Mann-Whitney test.

SECONDARY OUTCOMES:
Evaluation of CT perfusion parameters as predictive factors of response on baseline and on early follow-up | Through study completion, an average of 1 year
  Assessed using logistic regression

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No